CLINICAL TRIAL: NCT01151306
Title: The Cardiovascular and Inflammatory Effects of Statin Therapy in Patients With COPD
Brief Title: The Effect of Statins in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09105
Record Dates: First submitted 2010-06-21; First posted 2010-06-28 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Simvastatin; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactose tablet (Placebo Comparator)
  Interventions: Drug: Lactose tablet
- Simvastatin 20mg (Active Comparator)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 20mg once daily (in the evening) for 6 weeks
  Arms: Simvastatin 20mg
Drug: Lactose tablet — One tablet taken each evening for 6 weeks
  Arms: Lactose tablet

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a condition of the lungs which results in breathing difficulties due to the lungs becoming inflamed and the airways narrowed. Current treatments have focused on opening up the narrowed airways but, in addition, we know there is increased inflammation in the blood and these patients are at increased risk of heart disease. Statins, simvastatin being one of them, are drugs used to lower cholesterol in the blood but may also reduce inflammation and lower the risk of heart disease. This study will explore whether simvastatin reduces one of the risk factors in patients with COPD in a short term proof of principle study. The key purpose is to determine whether simvastatin improves the pressure and stiffness of the main blood vessels namely the arterial stiffness measure of aortic pulse wave velocity (PWV). In parallel, we will describe changes in airways and / or blood inflammation and change in breathing ability

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 45-80 years;
* Confirmed COPD: FEV1 30-80% predicted, FEV1/FVC<0.7, salbutamol reversibility <12%, supportive smoking history
* If female of childbearing potential, have a negative serum pregnancy test at screening and use a medically acceptable form of contraception starting at screening and continuing throughout the study (defined as an oral contraceptive, or barrier method combined with a spermicide)
* Able to attend for regular clinic appointments
* In opinion of investigator, the patient will be able to comply with the requirements of the protocol
* Provide written informed consent.

Exclusion Criteria:

* Known hypersensitivity to or side effects relating to previous statin treatment, or current therapy which includes a statin, ezetimibe or fibrate
* Clinically significant liver function abnormality; alcohol excess
* Hypercholesterolaemia > or equal to 6.5mmol/L
* Females who are pregnant, breast feeding, or at risk of pregnancy and not using a medically acceptable form of contraception.
* Any condition judged by investigator that would cause the study to be detrimental to patient.
* Conditions: rheumatoid disease/other collagen vascular disease requiring therapy; diabetes mellitus; untreated hypothyroidism; inflammatory bowel disease; other respiratory disease; known alpha 1 antitrypsin deficiency; malignancy; documented history of ischaemic heart disease (IHD); cor pulmonale or known congestive heart failure; patients planning to undergo elective surgery during the study period.
* Exacerbation in the last 4 weeks.
* Significant hypoxia (PaO2 <7.3kPa)
* Known lactose intolerance.
* Therapies: oral prednisolone for more than 1 week in the last 6 months; disease modifying drugs (Gold/ sulphasalazine etc); weight losing drugs; concomitant use of warfarin, cyclosporine; concomitant administration of potent CYP3A4 inhibitors (e.g. itraconazole, ketoconazole, HIV protease inhibitors, erythromycin, clarithromycin, telithromycin and nefazodone). Use of any investigational drug within four weeks of the baseline visit.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in arterial stiffness as measured by aortic pulse wave velocity (PWV) over study period | Week 0 (start) and week 6 (end)
  Aortic Pulse wave velocity (Sphygmocor, Atcor)

SECONDARY OUTCOMES:
Change in Circulating Inflammatory Mediators over study period | Week 0 (Start) and week 6 (End)
Change in distance (metres)walked on 6 minute walking test | week 0 (start) and week 6 (end)
  together with pre- and post-walk oxygen saturations
Change in blood total cholesterol, triglycerides, HDL and LDL over study period | week 0 (Start) and week 6 (End)
Change in airway inflammatory markers (differential cell count, exhaled nitric oxide and airway cytokines) over study period | week 0 and week 6
Change in lung function: Spirometry - forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) | week 0 (Start) and week 6 (End)
Change on blood pressure over study period | Week 0 (start) and Week 6 (end)
Change in Liver function tests | Week 0 (start) and Week 6 (End)
Change in creatine phosphokinase (CPK) over study period | Week 0 (start) and Week 6(End)
Change in Handgrip strength over study period | Week 0 (start) and Week 6 (end)
Change in blood desmosine over study period | Week 0 (Start) and Week 6 (end)
Change in circulating matrix metalloproteinase over study period | Week 0 (start) and Week 6 (end)
Baseline arterial stiffness (aortic pulse wave velocity) | Week 0
Baseline airway (differential cell count, exhaled nitric oxide and cytokines)and circulating inflammatory status (cytokines) | Week 0
Baseline matrix metalloproteinase in airway and blood | Week 0

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Respiratory Biomedical Research Unit, Nottingham, United Kingdom

REFERENCES:
- [Derived] John ME, Cockcroft JR, McKeever TM, Coward WR, Shale DJ, Johnson SR, Thornton JG, Harrison TW, Knox AJ, Bolton CE. Cardiovascular and inflammatory effects of simvastatin therapy in patients with COPD: a randomized controlled trial. Int J Chron Obstruct Pulmon Dis. 2015 Jan 29;10:211-21. doi: 10.2147/COPD.S76061. eCollection 2015. PMID 25673981